CLINICAL TRIAL: NCT05449158
Title: Effects of Left Atrial Pressure-guided Ventricular Rate Regulation on Cardiac Function in Patients Therapy With Atrioventricular Node Ablation Combined With Left Bundle Branch Pacing
Brief Title: The Relationship Between Left Atrial Pressure and Cardiac Function After Atrioventricular Node Ablation
Acronym: LAP-TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director of Cardiology, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAP-TOP
Record Dates: First submitted 2022-06-28; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation;; atrioventricular node ablation;; left bundle branch pacing
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAP Group (Experimental): Control of left atrial pressure changes by adjusting pacemaker frequency
  Interventions: Procedure: left atrial pressure regulation
- Control Group (No Intervention): General pacemaker rate setting

INTERVENTIONS:
Procedure: left atrial pressure regulation — For patients after atrioventricular node ablation combined with left atrial appendage closure, the regulation of left atrial pressure can be controlled by adjusting the frequency of pacemaker.
  Arms: LAP Group

SUMMARY:
Effects of left atrial pressure-guided ventricular rate changes on cardiac function after atrioventricular node ablation combined with left bundle branch pacing

DETAILED DESCRIPTION:
Effects of left atrial pressure-guided ventricular rate changes on cardiac function after atrioventricular node ablation combined with left bundle branch pacing. For patients with non-valvular atrial fibrillation who received atrioventricular node ablation combined with left bundle branch pacing in our hospital, a left atrial pressure catheter was used to monitor atrial pressure during the operation, and a lower average atrial pressure was obtained by adjusting the pacing frequency of the pacemaker. In a randomized controlled manner, the postoperative echocardiography, cardiothoracic ratio, cardiac function, etc. were compared between patients without atrial pressure monitoring and those who received atrial pressure adjustment, in order to clarify the effect of left atrial pressure-guided ventricular rate adjustment on atrioventricular node ablation combined with left bundle Benefit of pacing patients.

ELIGIBILITY:
Inclusion Criteria:

18-85 years old atrial fibrillation patients

Exclusion Criteria:

There is a history of pacemaker implantation; patients after coronary artery bypass grafting; severe coronary stenosis or occlusion cannot be treated with reperfusion;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
EF% | 1-year
  aortic vestibular ejection fraction

SECONDARY OUTCOMES:
cardiovascular all-cause mortality | 1week
  Proportion of patients dying from cardiovascular causes
Hospitalizations for heart failure | 1 years
  Hospitalizations for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, Ph.D, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Jun Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: After the research results are published；2 years；
Access Criteria: open
URL: http://www.chictr.org.cn/index.aspx